CLINICAL TRIAL: NCT02958644
Title: Effect of Synbiotic Supplement on the Body Mass Index of Participants With Severe Obesity
Acronym: Synbiotic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Dona Helena (Other)
Responsible Party: Principal Investigator, Marilyn Gonçalves Ferreira Kuntz, Principal Investigator, Hospital Dona Helena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDonaHelena
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Obesity Class III
Keywords: synbiotic; obesity; body mass index; microbiota
MeSH Terms: conditions — Obesity | interventions — Synbiotics; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotics (Experimental): Synbiotics - 12g / day fructo-oligosaccharide and probiotics supplemented orally for 90 days.
  Interventions: Dietary Supplement: Synbiotics
- Placebo (Placebo Comparator): Placebo - polydextrose 12g /day supplemented orally for 90 days.
  The study supplements are packed in identical envelopes containing either 12g of oral powder fructo-oligosaccharide and probiotics or placebo to be diluted in water. The powder and the solution were identical in appearance, taste, and smell.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotics — 12g / day synbiotics (fructo-oligosaccharide and probiotics) supplemented orally for 90 days
  Other Names: Fructo-oligosaccharide and probiotics
  Arms: Synbiotics
Dietary Supplement: Placebo — 12g / day placebo (polydextrose) supplemented orally for 90 days
  Arms: Placebo

SUMMARY:
Obese patients have a high level of intestinal microflora imbalance, with serious consequences such as loss of digestive function. Potential mediators of intestinal microbiota are prebiotics, supplements considered safe because they are naturally contained in food and human microbiota. Probiotics are living bacteria which are found in the normal gut microbiota. Synbiotics are combinations of both prebiotics and probiotics. Their use has been studied as a new therapeutic approach for the regulation of intestinal microbiota in various situations of disease, including severe obesity.

This is a double-blind, placebo-controlled, randomized clinical trial to assess the effect of synbiotic supplementation (fructo-oligosaccharide and probiotic - 12 g / day) on body mass index in participants with obesity class III, with follow up of 90 days.

DETAILED DESCRIPTION:
Obesity has been discussed as one of the major diseases that require scientific and technological innovations for its control is obesity and studies indicate that microbiota of obese patients have a high level of intestinal microflora imbalance, with serious consequences such as loss of digestive function and the combination of toxins to protein.

Potential mediators of intestinal microbiota are prebiotics, probiotics and synbiotics, supplements considered safe because they are naturally contained in food and human microbiota. Its use has been studied as a new therapeutic approach for the regulation of intestinal microbiota in various situations of disease, including in severe obesity.

This study aims to analyze the effect of synbiotics supplementation on body mass index in participants diagnosed with morbid obesity. The methodology used is the randomized clinical trial, placebo-controlled with blinding of patients, healthcare staff and outcome assessors, with follow-up of 90 days.

Patients will be randomized into two groups: control group to receive placebo (polydextrose - 12 g / day) and synbiotic group - group supplemented with synbiotic (fructo-oligosaccharide and probiotics - 12 g / day). Probiotics are: Lactobacillus acidophilus; Lactobacillus rhamnosus; Lactobacillus paracasei; Bifïdobacterium lactis.

At the moments proposed in this study, will be conducted assessments of food intake, nutritional status and metabolic / inflammatory parameters (body mass index, high-sensitivity C-reactive protein, albumin, triglycerides, total cholesterol, HDL-cholesterol and LDL-cholesterol, fasting blood glucose, glycated hemoglobin, fasting insulin, weight, height).

ELIGIBILITY:
Inclusion Criteria:

* Obesity class III (body mass index ≥40kg/m2)

Exclusion Criteria:

* Current use of prebiotics and probiotics or use in the last three months
* Intolerance to prebiotics and probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 90 days

SECONDARY OUTCOMES:
Plasma C-reactive protein | 90 days
Total cholesterol | 90 days
Plasma LDL-cholesterol | 90 days
Plasma HDL-cholesterol | 90 days
Plasma triglycerides | 90 days
Blood glucose | 90 days
  Fasting blood glucose
Glycated hemoglobin | 90 days
Plasma insulin | 90 days
Arterial blood pressure | 90 days
  Systolic and diastolic arterial blood pressure
Interleucin I-ß | 90 days
Interleucin 6 | 90 days
Albumin | 90 days
Tumoral Necrose Factor (TNF-α) | 90 days
Adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn G Ferreira, PhD, Study Chair — Hospital Dona Helena
Locations (3):
- Brazil (3):
  - Hospital Dona Helena, Joinville, Santa Catarina
  - Hospital Regional Hans Dieter Schmidt, Joinville, Santa Catarina
  - Hospital do Coração, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
We will share the database containing de-identified individual participant data, data dictionary documentation, statistical analysis plan, and analysis code. Beginning 6 months following article publication, the trial steering committee will evaluate proposals of studies accompanied by a statistical analysis plan and may grant access to the data for approved proposals.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months following article publication.
Access Criteria: The trial steering committee will evaluate proposals of studies accompanied by a statistical analysis plan and may grant access to the data for approved proposals.